CLINICAL TRIAL: NCT01944475
Title: Follow-up of Girls With Premature Thelarche and Precocious Puberty: a Clinical and Paraclinical Study of Girls With Thelarche and Healthy Controls
Brief Title: Follow-up of Girls With Premature Thelarche and Precocious Puberty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Mia Elbek Sømod, Research assistamt, University of Aarhus
Other Study IDs: 1-10-72-186-13
Record Dates: First submitted 2013-09-05; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Precocious Puberty; Excess; Development, Breast
Keywords: Precocious puberty; Premature thelarche; Tanner-stage; GnRH-test
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Observational Model: Case-Only
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — GnRH test, p-estrogen, p-testosterone , p-SHBG, p- androstenedione, p-dihydroandrostendion, p-inhibin B, p-thyroid parameters, ultrasound examination of the genitalia interna and a blood sample for studies of polymorphism in the estrogen receptor gene and aromatase enzyme gene.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Precocious puberty - the onset of signs of puberty before 8 years of age in girls - is be physically and emotionally devastating for kids and is sometimes caused by an underlying and medical condition. One sign of precocious puberty in small girls is breast development (thelarche). This can persist without other physical changes of puberty, it may continue into precocious puberty, or it may disappear. This project will improve the diagnostics of precocious puberty in girls and improve our ability to identify which girls with thelarche, who will develop precocious puberty and need medical treatment.

DETAILED DESCRIPTION:
The purpose of the study is

1. To conduct an epidemiological study in which characteristics of 0-6 year-old girls with either premature thelarche or precocious puberty are described (as specified below)
2. To conduct a clinical and para-clinical re-examination of the before-mentioned (1))0-6 year-old girls
3. To compare the clinical and paraclinical parameters in point 1) mentioned 0-6 year-old girls with a control group of children at the same age, whiteout thelarche and precocious puberty. (Local Ethics Committee has approved the study of the control group, case number 1-10-72-631-12.)

The study includes a chart review of registered 0-6 year-old girls diagnosed with premature thelarche or precocious puberty from 1998 and until today at Dept. of Pediatrics A, AUH Skejby. The cohort has not earlier been examined and the number of girls in the cohort is estimated from our clinical experience with this patient group to be about 50 in total. The following characteristics from the patients records will be registered in a database:

Age at diagnosis, anthropometry (height and weight), Tanner stage - breast, Tanner stage - pubic hair, GnRH test (LH and FSH response), thyroid parameters, estrogen, prolactin, 17OHP, androstenedione, dihydroepiandrosteron (DHEA), testosterone, inhibin B, SHBG, AFP, kisspeptin, human chorionic gonadotropin (HCG), bone age, MRI of the cerebrum, US of internal genitalia, and exposures to environmental chemicals known to affect secondary sex characteristics.

The database will be developed in the program Access. The results will be reported as mean and standard deviation and minimum and maximum values for each age group by Tanner stage, if the data are normally distributed. Non-normally distributed data will be given as median and confidence intervals as well as minimum and maximum values for each Tanner stage. Data for previously studied children with suspected precocious puberty, will be reported in the same way. Statistical comparison between the groups will be made with u-paired t-test or equivalent non-parametric test, if the data is not normally distributed.

The Data Unit at Aarhus University Hospital, Skejby, identifies 0-6 year-old girls with diagnoses premature thelarche or precocious puberty in 1998 and onwards. Girls below 8 years of age at baseline of the project (1st of September 2013) will be contacted and requested to participate in a re-examination.

The follow-up is a clinical and paraclinical re-examination, where the following parameters are measured: anthropometry (height and weight), skinfold thickness, Tanner stage, bone age, GnRH test, p-estrogen, p-testosterone , p-SHBG, p- androstenedione, p-dihydroandrostendion, p-inhibin B, p-thyroid parameters, ultrasound examination of the genitalia interna and a blood sample for studies of polymorphism in the estrogen receptor gene and aromatase enzyme gene.

If the girls are unable or unwilling to attend the reexamination, they are requested to fill out a questionnaire instead as follows:

* name, social security number, date of completion the questionnaire
* current height, current weight, birth weight, origin
* date of onset of puberty if started, current pubertal development, menarche
* diseases/admissions

Regarding the mother:

- age at menarche, medicine during pregnancy/breastfeeding, diet during pregnancy/breastfeeding, use of cosmetics /cream/shampoo during pregnancy,

Regarding the family:

- others with early breast development/early puberty

The project is conducted at Dept. of Pediatrics A, Aarhus University Hospital, Skejby, Skejbygårdsvej 100, 8200 Aarhus N. The other pediatric wards in the Region of Midtjylland (located in Randers, Viborg and Herning) will be included in the project if they prefer to participate.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of precocious puberty or premature thelarche
* 0-6 year old girls at time of diagnosis for the medical record review
* 0-8 year old girls at baseline for the re-examination

Exclusion Criteria:

-

Max Age: 8 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: 0-6 year old girls diagnosed with premature thelarche or precocious puberty from 1998 to today at the Children's Section A, AUH, Skejby. Girls who are 8 years old or under at baseline (1st of september) will be contacted and asked to participate in a clinical and paraclinical re-examination.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Tanner stage (breast and pubic hair) | Up till age 21.0 years

SECONDARY OUTCOMES:
weight | up till age 21.0 years
height | Up till age 21.0 years
Bone age | Up till age 21.0 years
LH-peak after GnRH-test | Up till age 21.0 years
Hormones (estrogen, prolactin, 17OHP, androstrendion, DHEA, testosterone, inhibin B, SHBG, AFP, kisspeptin, HCG, thyroid hormones) | Up till age 21.0 years
Ultrasound of the internal genitalia | Up till age 21.0 years

OTHER OUTCOMES:
Exposure | Up till age 21.0 years

CONTACTS AND LOCATIONS:
Overall Officials: Niels H. Birkebæk, MD PhD, Principal Investigator — Børneafdeling A, AUH, Skejby; Esben T. Vestergaard, MD, PhD, Principal Investigator — Børneafdeling A, AUH, Skejby; Kurt Kristensen, MD, PhD, Principal Investigator — Børneafdeling A, AUH, Skejby; Mia E. Sømod, Stud.med, Principal Investigator — Børneafdeligen A, AUH, Skejby
Locations (1):
- Børneafdelingen A, AUH, Skejby, Aarhus N, Denmark

REFERENCES:
- [Background] Carel JC, Leger J. Clinical practice. Precocious puberty. N Engl J Med. 2008 May 29;358(22):2366-77. doi: 10.1056/NEJMcp0800459. No abstract available. PMID 18509122
- [Background] Carel JC, Lahlou N, Roger M, Chaussain JL. Precocious puberty and statural growth. Hum Reprod Update. 2004 Mar-Apr;10(2):135-47. doi: 10.1093/humupd/dmh012. PMID 15073143
- [Background] Tremblay L, Frigon JY. Precocious puberty in adolescent girls: a biomarker of later psychosocial adjustment problems. Child Psychiatry Hum Dev. 2005 Fall;36(1):73-94. doi: 10.1007/s10578-004-3489-2. PMID 16049645
- [Background] Michaud PA, Suris JC, Deppen A. Gender-related psychological and behavioural correlates of pubertal timing in a national sample of Swiss adolescents. Mol Cell Endocrinol. 2006 Jul 25;254-255:172-8. doi: 10.1016/j.mce.2006.04.037. Epub 2006 Jun 27. PMID 16806671
- [Background] Herman-Giddens ME, Slora EJ, Wasserman RC, Bourdony CJ, Bhapkar MV, Koch GG, Hasemeier CM. Secondary sexual characteristics and menses in young girls seen in office practice: a study from the Pediatric Research in Office Settings network. Pediatrics. 1997 Apr;99(4):505-12. doi: 10.1542/peds.99.4.505. PMID 9093289
- [Background] Teilmann G, Pedersen CB, Jensen TK, Skakkebaek NE, Juul A. Prevalence and incidence of precocious pubertal development in Denmark: an epidemiologic study based on national registries. Pediatrics. 2005 Dec;116(6):1323-8. doi: 10.1542/peds.2005-0012. PMID 16322154
- [Background] Houk CP, Kunselman AR, Lee PA. The diagnostic value of a brief GnRH analogue stimulation test in girls with central precocious puberty: a single 30-minute post-stimulation LH sample is adequate. J Pediatr Endocrinol Metab. 2008 Dec;21(12):1113-8. doi: 10.1515/jpem.2008.21.12.1113. PMID 19189683
- [Background] Curfman AL, Reljanovic SM, McNelis KM, Dong TT, Lewis SA, Jackson LW, Cromer BA. Premature thelarche in infants and toddlers: prevalence, natural history and environmental determinants. J Pediatr Adolesc Gynecol. 2011 Dec;24(6):338-41. doi: 10.1016/j.jpag.2011.01.003. PMID 22099730
- [Background] Atay Z, Turan S, Guran T, Furman A, Bereket A. The prevalence and risk factors of premature thelarche and pubarche in 4- to 8-year-old girls. Acta Paediatr. 2012 Feb;101(2):e71-5. doi: 10.1111/j.1651-2227.2011.02444.x. Epub 2011 Sep 23. PMID 21854448
- [Background] de Vries L, Guz-Mark A, Lazar L, Reches A, Phillip M. Premature thelarche: age at presentation affects clinical course but not clinical characteristics or risk to progress to precocious puberty. J Pediatr. 2010 Mar;156(3):466-71. doi: 10.1016/j.jpeds.2009.09.071. Epub 2009 Nov 14. PMID 19914634